CLINICAL TRIAL: NCT02579460
Title: Reflux-Induced Oxidative Stress in Barrett's Esophagus: Response, Repair, and Epithelial-Mesenchymal-Transition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dallas VA Medical Center (U.S. Federal Agency)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Stuart Spechler, Professor of Medicine, Dallas VA Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 15-022; 1R01DK103598-01A1 (NIH)
Record Dates: First submitted 2015-10-14; First posted 2015-10-19 (Estimated); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Barrett's Esophagus; Gastroesophageal Reflux Disease
Keywords: Barrett's esophagus; Gastroesophageal Reflux Disease
MeSH Terms: conditions — Barrett Esophagus; Gastroesophageal Reflux

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Barrett's esophagus patients (Experimental): Patients with Barrett's Esophagus will be enrolled. The intervention is cessation of acid-suppressing medications. Biopsies will be taken during endoscopy at Day 0, 7, and 14.
  Interventions: Other: Cessation of Acid Suppressing Medications

INTERVENTIONS:
Other: Cessation of Acid Suppressing Medications — Acid suppressing medications are stopped for all participants the day after baseline assessment. Subsequent evaluations are performed while the participant is not on acid-suppressing medications. Endoscopy with biopsies will be performed in all patients on day 0, 7, and 14.

SUMMARY:
The purpose of this study is to elucidate mechanisms whereby oxidative stress induced by acute reflux esophagitis: 1) activates p38 to regulate proteins that control the G1/S cell cycle checkpoint, and 2) activates HIFs (hypoxia inducible factors) to cause autocrine VEGF (vascular endothelial growth factor) signaling that triggers the EMT (epithelial-mesenchymal-transition) program in Barrett's esophagus.

DETAILED DESCRIPTION:
Gastroesophageal reflux disease (GERD) and its complication, Barrett's esophagus (BE), are risk factors for esophageal adenocarcinoma. In BE, GERD causes inflammation with oxidative DNA damage and genomic instability that contributes to carcinogenesis. In BE, one response to oxidative stress is p38 pathway activation, which might protect against cancer development by initiating G1 arrest and enabling repair of DNA damage. Inflammation and oxidative stress also might induce epithelial-mesenchymal transition (EMT), the process in which epithelial cells acquire mesenchymal characteristics including the ability to migrate. This study will elucidate mechanisms whereby the oxidative stress of acute reflux esophagitis in BE activates p38 to regulate proteins controlling the G1/S cell cycle checkpoint, and activates HIFs to cause autocrine vascular endothelial growth factor (VEGF) signaling that triggers the EMT program.

ELIGIBILITY:
Inclusion Criteria:

* U.S. Veteran
* Barrett's Esophagus

Exclusion Criteria:

* Inability to provide informed consent
* Pregnancy or breastfeeding
* Esophageal varices
* Warfarin use
* Coagulopathy that precludes safe biopsy of the esophagus
* Comorbidity that precludes safe participation in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change in esophageal mucosal inflammation using histopathological assessment from baseline to 14 days | day 0, day 7, and day 14
  Inflammation of the esophageal mucosa will be measured at baseline, 7 days, and at 14 days. Esophageal mucosal inflammation will be measured using esophageal mucosal biopsy specimens, and histopatholgical grading. Mucosal infiltration with inflammatory cells (neutrophils, eosinophils, and lymphocytes) will be measured.

SECONDARY OUTCOMES:
change in p38 pathway from baseline to 14 days | day 0, day 7, and day 14
  p38 and components of the p38 pathway will be measured in the esophageal mucosa at baseline, 7 days, and at 14 days
change in phosoho-p38 from baseline to 14 days | day 0, day 7, and day 14
  phospho-p38 will be measured in the esophageal mucosa at baseline, day 7, and at day 14
Show oxidative DNA damage associated with p38 activation | day 0, day 7, and day 14
  OxiSelect Oxidative DNA Damage ELISA assay of Barrett's mucosa at baseline, day 7, and day 14
change in VEGF from baseline to 14 days | day 0, day 7, and day 14
  VEGF will be measured in the esophageal mucosa at baseline, 7 days, and at day 14
change in APE-1 from baseline to 14 days | day 0, day 7, and day 14
  APE-1 will be measured in the esophageal mucosa at baseline, day 7, and at day 14
change in NPM1 from baseline to 14 days | day 0, day 7, and day 14
  NPM-1 will be measured in the esophageal mucosa at baseline, day 7, and at day 14
change in phospho-NPM1 from baseline to 14 days | day 0, day 7, and day 14
  phospho-NPM1 will be measured in the esophageal mucosa at baseline, day 7, and at day 14
change in miRNA expression from baseline to 14 days | day 0, day 7, and day 14
  miRNAs will be measured in the esophageal mucosa and in exosomes isolated from the blood at baseline, day 7, and day 14
change in HIF expression from baseline to 14 days | day 0, day 7, and day 14
  HIF expression will be measured in the esophageal mucosa at baseline, day 7, and day 14

CONTACTS AND LOCATIONS:
Overall Officials: Stuart J Spechler, MD, Principal Investigator — Dallas VA Medical Center
Locations (1):
- Dallas VA Medical Center, Dallas, Texas, United States

REFERENCES:
- [Derived] Zhang Q, Dunbar KB, Odze RD, Agoston AT, Wang X, Su T, Nguyen AD, Zhang X, Spechler SJ, Souza RF. Hypoxia-inducible factor-1alpha mediates reflux-induced epithelial-mesenchymal plasticity in Barrett's oesophagus patients. Gut. 2024 Jul 11;73(8):1269-1279. doi: 10.1136/gutjnl-2023-331467. PMID 38641363